CLINICAL TRIAL: NCT06040970
Title: A Single-Center, Open-Label, Single-Arm, Phase I Study With Dose Expansion Cohort of Sacituzumab Govitecan in Combination With Cisplatin in Platinum Sensitive Recurrent Ovarian and Endometrial Cancer
Brief Title: Sacituzumab Govitecan in Combination With Cisplatin in Platinum Sensitive Recurrent Ovarian and Endometrial Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Amy Tiersten, MD. Professor of Medicine (Hematology and Medical Oncology) Clinical Director, Breast Medical Oncology, Dubin Breast Center, Icahn School of Medicine at Mount Sinai
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY-23-00832
Record Dates: First submitted 2023-09-05; First posted 2023-09-18 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Ovarian Cancer; Malignant Neoplasm of Uterus
MeSH Terms: conditions — Ovarian Neoplasms; Uterine Neoplasms | interventions — sacituzumab govitecan; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Ovarian cancer Cohort (Experimental): DEC 3+3 dose expansion of Sacituzumab Govitecan in Combination with Cisplatin
  Interventions: Drug: Sacituzumab; Drug: Cisplatin
- Endometrial cancer Cohort (Experimental): DEC 3+3 dose expansion of Sacituzumab Govitecan in Combination with Cisplatin
  Interventions: Drug: Sacituzumab; Drug: Cisplatin

INTERVENTIONS:
Drug: Sacituzumab — Dose 0: Sacituzumab govitecan 7.5 mg/kg
  Dose -1: Sacituzumab govitecan 5 mg/kg
  Other Names: Sacituzumab Govitecan
Drug: Cisplatin — Cisplatin 70 mg/m2 IV

SUMMARY:
This is an open-label, Phase 1 study with a dose expansion cohort of Sacituzumab Govitecan in Combination with Cisplatin in Platinum Sensitive Recurrent Ovarian and Endometrial Cancer. The goal of the study is to determine the optimal dose of sacituzumab govitecan for use in combination with cisplatin for treatment of epithelial ovarian and endometrial cancers.

DETAILED DESCRIPTION:
This is an open-label, Phase 1 study with a dose expansion cohort (DEC), conducted in two separate disease groups (ovarian and endometrial cancer). The primary objective of the study is to determine the optimal dose of sacituzumab govitecan for use in combination with cisplatin for treatment of epithelial ovarian and endometrial cancers.

For each disease group, there will be a safety run-in phase utilizing a 3+3 design with a de-escalated dose level if the starting dose shows toxicity and an expansion cohort to evaluate the preliminary efficacy and tolerability of the experimental regimen. The dose expansion cohort will consist of 14 patients in the ovarian cohort and 12 patients in the endometrial cohort with an additional 2 patients in each cohort to account for potential patient replacement. This will yield a total sample size of 22-28 patients in the ovarian cancer cohort and a total sample size of 20-26 patients in the endometrial cancer cohort.

Phase 1, Safety Run-in with Dose De-escalation Scheme:

Dose Level 0, starting level: Sacituzumab govitecan 7.5 mg/kg + Cisplatin 70 mg/m2 IV Dose -1: Sacituzumab govitecan 7.5 mg/kg + Cisplatin 70 mg/m2 IV In this stage, a minimum of 6 patients and a maximum of 12 patients will be required.

The recommended dose expansion cohort (DEC) dose is defined as the highest dose at which no more than 1 out of 6 patients experience a Dose-Limiting Toxicity (DLT)

Phase 2, Dose Expansion Cohort:

Sacituzumab govitecan 5-7.5 mg/kg IV (depending on phase I result) + Cisplatin 70 mg/m2 IV.

Drug product administration will continue until progressive disease (PD), unacceptable toxicity, or death.

The primary endpoint of the safety run-in phase is to determine the recommended DEC dose of Sacituzumab in combination with a fixed schedule of cisplatin in patients with ovarian and endometrial cancers. In the safety run-in phase, the assessment of dose limiting toxicity (DLT) will be performed standard 3 + 3 design rules. The recommended DEC dose is defined as the highest dose of Sacituzumab in combination with Cisplatin at the fixed dose of 70 mg/m2 at which no more than 1 out of 6 patients experience DLT within the first cycle of therapy.

The DEC is designed to indicate proof of concept regarding the overall response rate (ORR) and safety of the combination of sacituzumab with cisplatin at the dose established in the safety run-in phase of the study. Once the recommended DEC dose for sacituzumab and cisplatin combination has been established for each disease cohort, an additional 14 patients will be enrolled for the ovarian group and 12 patients for the endometrial group. An additional 2 patients will be added to each cohort to account for potential patient replacement for a total of 42-54 evaluable patients.

ELIGIBILITY:
Eligibility waivers are not permitted. Subjects must meet all of the inclusion and exclusion criteria to be registered to the study. Study treatment may not begin until a subject is registered.

Inclusion Criteria:

* Pathologic (histology or cytology) confirmed diagnosis of epithelial ovarian cancer or endometrial cancer
* Radiographic evidence of recurrent epithelial ovarian cancer (ovarian, fallopian tube, or primary peritoneal cancer) or endometrial cancer that is "platinum-sensitive," defined as progression of disease beyond 6 months from the last dose of platinum-based chemotherapy
* Female, age ≥ 18 years
* World Health Organization (WHO) performance status 0-1 with no deterioration over the previous 2 weeks and minimum life expectancy of 12 weeks
* Patient has measurable disease (at least one lesion that can be accurately assessed repeatedly by CT) as evidenced on pre-treatment baseline CT of Chest/Abdomen/Pelvis or PET/CT, or evaluable disease
* Adequate hematologic counts, as defined below, without transfusion or growth factor support within 2 weeks of study drug initiation:

  * Hemoglobin ≥ 8.5 g/dL
  * Absolute neutrophil count ≥ 1500/mm3
  * Platelets ≥ 100,000/μL
* Adequate organ function as defined below:

  * Total bilirubin ≤ 1.5 ULN
  * AST(SGOT)/ALT(SPGT) ≤ 2.5x ULN or ≤ 5 x ULN if known liver metastases
  * Serum albumin > 3 g/dL
  * Creatinine clearance ≥ 50 mL/min per the Cockcroft-Gault equation
* Women of childbearing potential must agree to use adequate contraception prior to study entry, for the duration of study participation, and for 6 months following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

  o A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
  * Has not undergone a hysterectomy or bilateral oophorectomy; or
  * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

Treatment with any of the following:

* Any investigational agents or study drugs from a previous clinical study within 28 days or 5 half-lives (whichever is longer) of the first dose of study treatment
* Any other chemotherapy, immunotherapy or anticancer agents within 14 days of the first dose of study treatment
* Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study treatment
* Radiotherapy with a wide field of radiation within 4 weeks or radiotherapy with a limited field of radiation for palliation within 2 weeks of the first dose of study treatment
* With the exception of alopecia, any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) grade 1 at the time of starting study treatment
* As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including active bleeding diatheses, or uncontrolled infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV). Screening for chronic conditions is not required.
* Known or severe (Grade 3 or higher) hypersensitivity to SG and/or cisplatin, their metabolites, or formulation excipients
* Peripheral neuropathy grade 2 or greater
* Refractory nausea and vomiting, chronic gastrointestinal diseases
* Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Women of childbearing potential unwilling to use effective contraception during study until conclusion of 6-month post-treatment evaluation period
* Known history of unstable angina, MI, or CHF present within 6 months of randomization or clinically significant cardiac arrhythmia (other than stable atrial fibrillation) requiring anti-arrhythmia therapy
* Known history of clinically significant active COPD, or other moderate-to-severe chronic respiratory illness present within 6 months of enrollment.
* Prior history of clinically significant bleeding, intestinal obstruction, or GI perforation within 6 months of enrollment.
* Other concurrent medical or psychiatric conditions that, in the Investigator's opinion, may be likely to confound study interpretation or prevent completion of study procedures and follow-up examinations.
* Prior therapy with sacituzumab govitecan, irinotecan, Trop-2-directed antibody drug conjugate, or any topoisomerase I-containing antibody-drug conjugates at any time for early stage disease
* Have active chronic inflammatory bowel disease (ulcerative colitis, Crohn's disease) or GI perforation within 6 months of enrollment.
* Requirement for ongoing therapy with any prohibited medications
* Have known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they have stable CNS disease for ≥ 4 weeks prior to randomization and all neurologic symptoms have returned to baseline, have no evidence of new or enlarging brain metastases, and are taking 10 mg/day or less of prednisone or its equivalent. All participants with carcinomatous meningitis are excluded regardless of clinical stability.
* Have an active second malignancy. Participants with a history of malignancy that have been completely treated, with no evidence of active cancer for 3 years prior to randomization, or participants with surgically cured tumors with low risk of recurrence (e.g., nonmelanoma skin cancer, histologically confirmed complete excision of carcinoma in situ, or similar) are allowed to enroll.
* Use of any live vaccine against infectious diseases within 30 days of the first dose of study drugs.
* Have an active serious infection requiring systemic antimicrobial therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 54 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (DLT) at the maximum tolerated dose (MTD) for the Safety Run-In Phase | within the first cycle of therapy (each cycle = 21 days)
  Safety Run-In Phase: The primary endpoint of the safety run-in phase is to determine DLT and the recommended DEC dose of sacituzumab govitecan in combination with a fixed schedule of cisplatin in patients with ovarian and endometrial cancers. DLT is defined as any therapy-attributable adverse event (AE) requiring discontinuation of therapy within one cycle of combined therapy; specifically grade 3 or 4 non-hematologic toxicity and grade 4 hematologic toxicity events. These will be assessed via NCI's CTCAE v 5.0 toxicity criteria. DEC dose is defined as the highest dose at which no more than 1 out of 6 patients experience a DLT.
  All primary endpoints will be reported separately for each of the ovarian and endometrial cohorts.
Dose limiting toxicity (DLT) for the DEC Phase | within 1 cycle of therapy (each cycle = 21 days)
  A primary endpoint for the dose expansion cohort (DEC) phase of this study will be the DLT rate evaluated within 1 cycle of sacituzumab in combination with cisplatin.
  The DLT rate is defined as the proportion of patients in the safety population of the phase 1 and dose expansion cohort (DEC) phase of the study that experience at least 1 DLT within the first cycle of sacituzumab in combination with cisplatin treated at the maximum tolerated dose (MTD).
  DLT is defined as any therapy-attributable adverse event (AE) requiring discontinuation of therapy within one cycle of combined therapy; specifically grade 3 or 4 non-hematologic toxicity and grade 4 hematologic toxicity events. These will be assessed via NCI's CTCAE v 5.0 toxicity criteria.
  All primary endpoints will be reported separately for each of the ovarian and endometrial cohorts.
Overall Response Rate (ORR) | every 3 cycles (each cycle is 21 days)
  A primary endpoint for the dose expansion cohort (DEC) phase will be the ORR evaluated within 3 cycles of sacituzumab in combination with cisplatin in patients with platinum-sensitive recurrent epithelial ovarian cancer and endometrial cancer. This will be measured every 3 cycles (12 weeks +/- 1 week).
  The overall response rate is defined as the proportion of patients in the full analysis (FA) population treated at the MTD, in both the phase 1 and DEC phases of the study, whose cancer decreases in size on assessment (as measured by the sum of complete response (CR) and partial response (PR)). Disease status will be assessed based on RECIST 1.1 criteria for measurable and non-measurable disease.
  The Full Analysis (FA) population includes all patients who received at least one cycle of all study medications and had at least one valid post-baseline efficacy assessment.
  All primary endpoints will be reported separately for each of the ovarian and endometrial cohorts.

SECONDARY OUTCOMES:
Clinical Benefit Response (CBR) | 6 months
  For the entire cohort (Safety Run-In and Dose Expansion Cohort), CBR will be measured by the percentage of patients whose cancer shrinks or remains stable over the duration of the study. This will be measured as the sum of complete response (CR), partial response (PR), and stable disease (SD) for greater than or equal to 6 months. Disease status will be assessed based on RECIST 1.1 criteria for measurable and non-measurable disease.
  The analysis plan for all secondary endpoints will be conducted separately for each disease cohort (ovarian and endometrial).
Progression free survival (PFS) | 6 months
  For the entire cohort (Safety Run-In and Dose Expansion Cohort), 6-month progression free survival (PFS) is as defined as the time from the start of treatment until confirmed disease progression or death from any cause, whichever occurs first. Disease status will be assessed with comprehensive radiographic studies every 3 treatment cycles (12 weeks +/- 1 week), but the development of new signs or symptoms of disease in between scheduled evaluations may prompt off-schedule radiographic or non-radiographic evaluations. Disease status will be assessed based on RECIST 1.1 criteria for measurable and non-measurable disease.
  The analysis plan for all secondary endpoints will be conducted separately for each disease cohort (ovarian and endometrial).
Number of adverse events | 6 months
  For the entire cohort (Safety Run-In and Dose Expansion Cohort), the type, incidence, severity (as graded by the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] v5.0), seriousness and relationship to study medications of Adverse Events will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Tiersten, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai Division of Hematology and Medical Oncology
Locations (1):
- Icahn School of Medicine at Mount Sinai Division of Hematology and Medical Oncology, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
There are no plans to share individual participant data, supporting information, or biological samples that are collected as part of this study for future research, even if the participant's identity is removed. Data and samples will only be used to complete this study. If the results of this study are presented or reported in a publication, the participants will not be identified. All results will be kept confidential and will not be divulged without permission, except as required by law.

DOCUMENTS (1):
  • Informed Consent Form (2025-04-29): https://cdn.clinicaltrials.gov/large-docs/70/NCT06040970/ICF_000.pdf